CLINICAL TRIAL: NCT06372613
Title: What is the Level of Serum Leucine-rich α 2-glycoprotein (LRG) Which Predicts Histologic Remission in Patients With Ulcerative Colitis?
Brief Title: Association Between LRG and Histologic Remission in Ulcerative Colitis
Status: Recruiting | Type: Observational
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Digestive Disease Center, Showa Inan General Hospital
Other Study IDs: LRG&UC
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis in Histologic Remission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
We attempt to clarify the serum leucine-rich α 2-glycoprotein (LRG) level which can predict histologic remission in ulcerative colitis patients in this study. Colonoscopy with histology will be performed when histologic remission is predicted, irrespective of symptoms or serum LRG values. Serum LRG levels are analyzed by an enzyme-linked immunosorbent assay.

DETAILED DESCRIPTION:
Aim: Serum leucine-rich α 2-glycoprotein (LRG) may be a noninvasive biomarker for monitoring disease activity in patients with ulcerative colitis (UC). We attempt to clarify the LRG level which predicts histologic remission in UC patients in this study.

Methods: Patients with UC were consecutively enrolled with the measurement of serum LRG. Colonoscopy with histology is performed when histologic remission is predicted, irrespective of symptoms or serum LRG values. Serum LRG levels are analyzed by an enzyme-linked immunosorbent assay. For the evaluation of UC activity, clinical remission was defined as score 1 or 0 using the partial Mayo score and endoscopic remission was defined as score 0 using the Mayo endoscopic subscore. And histologic remission is defined as < grade 2 using Geboes score. We analyze the area under receiver operating characteristic (ROC) curves to evaluate the diagnostic ability of LRG for predicting histologic remission of UC.

ELIGIBILITY:
Inclusion Criteria:

* active UC patients

Exclusion Criteria:

* None

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Active UC patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Histologic remission of UC | 1 week
  Histologic remission is defined as < grade 2 using Geboes score.

SECONDARY OUTCOMES:
Endoscopic remission | 1 week
  Endoscopic remission is defined as score 0 using the Mayo endoscopic subscore.

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Japan